CLINICAL TRIAL: NCT02526940
Title: Impact of Pre- Antiretroviral Therapy (ART) Blood Cluster of Differentiation (CD)4+ T Cell Level on the Rectal Reservoir in Long-term HIV-1 Treated Men
Brief Title: Impact of Pre-ART Blood CD4+ T Cell Level on the Rectal Reservoir in Long-term HIV-1 Treated Men
Acronym: VIRECT
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 1308020
Record Dates: First submitted 2015-08-17; First posted 2015-08-18 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Human Immunodeficiency Virus
Keywords: Human Immunodeficiency Virus; HIV; HAART; Highly Active antiretroviral therapy; GALT; Gut Associated Lymphoid Tissue; reservoir; rectum
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood specimen and rectal biopsies
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- blood CD4 cells count < 200/mm3: patients with blood CD4 cells count at the time of initiation of HAART< 200/mm3.
  Six rectal biopsies and blood samples collected for each patient treated by HAART more than 1 year and less than 4 years
  Interventions: Procedure: rectal biopsies; Other: Blood samples
- blood CD4 cells count : 200 - 300/mm3: patients with blood CD4 cells count at the time of initiation of HAART between 200 and 300/mm3 Six rectal biopsies and blood samples collected for each patient treated by HAART more than 1 year and less than 4 years
  Interventions: Procedure: rectal biopsies; Other: Blood samples
- blood CD4 cells count >350/mm3: patients with blood CD4 cells count at the time of initiation of HAART> 350/mm3.
  Six rectal biopsies and blood samples collected for each patient treated by HAART more than 1 year and less than 4 years
  Interventions: Procedure: rectal biopsies; Other: Blood samples

INTERVENTIONS:
Procedure: rectal biopsies — 6 rectal biopsies
Other: Blood samples — Blood samples

SUMMARY:
Although combined antiretroviral therapy (cART) has dramatically improved quality of life and lifespan of HIV infected individuals, it still fails to eliminate viral reservoirs. The Gut Associated Lymphoid Tissue (GALT) is the largest reservoir of HIV-1, as it harbors most of HIV target cells as activated memory Cluster of differentiation (CD)4+/CCR5+ T cells. Intestinal T and B cells express α4β7 integrin, a gut mucosal homing receptor which binds to gp120 HIV-1 envelope facilitating the infection of intestinal T cells and the early establishment of the gut HIV reservoir. Intensive viral replication in the GALT leads to an early impairment of mucosal immunity, due to the severe CD4+ T cells depletion, that could be also explained by a lack of recruitment in the gut. Among T cells, interleukin-(IL-)17 secreting CD4+ T cells (Th17) are particularly depleted during HIV infection. This depletion could be associated with HIV progression since these cells play a crucial role in the maintenance of mucosal immunity. A dysbalance of the Th17/Treg ratio may reflect the loss of the intestinal epithelial barrier integrity. These damages are responsible for an increase in microbial translocation, which is associated with immune activation and progression to AIDS. Several recent studies have shown that cART initiation during acute or early HIV-1 infection reduces HIV DNA reservoir size and improves immune reconstitution in blood. Post-treatment controllers, who started long-term cART early after HIV infection, have very low levels of HIV DNA in peripheral blood mononuclear cells, similarly to elite controllers. Unlike most HIV-infected individuals, they maintain an undetectable plasmatic viral load after several years of cART interruption, suggesting that a weak reservoir is a prerequisite to achieve a functional cure. By extrapolation, it could be hypothesized that the gut viral reservoir is also decreased and that mucosal immunity is restored when cART is initiated during primary phase of infection. The gut viral reservoir begins to form within the first days after HIV exposure, and grows during acute HIV infection. Similarly, intestinal T cells are depleted very early after infection, due to high viral replication, host immune response and bystander effects. Most studies also concluded that long-term and optimal treatment can't fully restore mucosal immunity. These observations led us to study the impact of time of cART start on the size of viral reservoir and on immune reconstitution in the gut. For this, we analyzed the virological and immunological characteristics of the rectal HIV reservoir of long-term treated patients regarding their blood CD4+ T cells count at the time of cART initiation.

ELIGIBILITY:
Inclusion Criteria:

* Seropositive for HIV
* Under HAART since at least one and less than 4 years
* No blood HIV RNA rebound during the therapy
* Indication of Human Papilloma Virus (HPV) screening by anal rectoscopy
* Signature of the informed consent form

Exclusion Criteria:

* Patient under tutelage
* No signature of the informed consent form
* No CD4 cell count available at the time of HAART initiation
* One or several viral rebound(s) during therapy
* Coinfection by hepatitis B virus (HBV) or hepatitis C virus (HCV)
* Hemostasis disorders, anticoagulant therapy
* No medical indication of rectoscopy
* Inflammatory bowel disease
* No understanding of the protocol

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 3 groups of men elaborated on the basis of their blood CD4+ T cells count at the time of cART initiation: >350; 350-200; <200, respectively.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-05; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
HIV DNA load in rectal biopsies | day 1
  Comparison of HIV DNA load (copies/106 cells) in rectal biopsies between 3 groups of patients (10 per group) according to their blood CD4 cells count at the time of initiation of Highly Active Antiretroviral Therapy (HAART) : <200, 200-300 and >350/mm3

SECONDARY OUTCOMES:
HIV DNA load in blood peripheral blood mononuclear cell (PBMC) | Day 1
  Comparison of HIV DNA load (copies/106 cells) in blood PBMC between 3 groups of patients (10 per group) according to their blood CD4 cells count at the time of initiation of HAART : <200, 200-300 and >350/mm3
HIV RNA load in blood PBMC | Day 1
  Comparison of HIV RNA load (copies/106 cells) in blood PBMC between 3 groups of patients (10 per group) according to their blood CD4 cells count at the time of initiation of HAART : <200, 200-300 and >350/mm3
HIV RNA load in rectal biopsies | Day 1
  Comparison of HIV RNA load (copies/106 cells) in rectal biopsies between 3 groups of patients (10 per group) according to their blood CD4 cells count at the time of initiation of HAART : <200, 200-300 and >350/mm3
Cellular composition in rectal biopsies | Day 1
  Comparison of Cellular composition in rectal biopsies between 3 groups of patients (10 per group) according to their blood CD4 cells count at the time of initiation of HAART : <200, 200-300 and >350/mm3.
  Cellular composition is a outcome measure : expression of CD3, CD4, CD8, CD27, CD45, CCR5 by flow cytometry
Cellular composition in blood PBMC | Day 1
  Comparison of Cellular composition in blood PBMCbetween 3 groups of patients (10 per group) according to their blood CD4 cells count at the time of initiation of HAART : <200, 200-300 and >350/mm3.
  Cellular composition is a outcome measure : expression of CD3, CD4, CD8, CD27, CD45, CCR5 by flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Frederic LUCHT, PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-ETIENNE, Saint-Etienne, France